CLINICAL TRIAL: NCT02742194
Title: Double-blind Placebo-controlled Clinical Trial of Ginger (Zingiber Officinale) Addition in the Obesity Treatment and Improvement Behavioral Profile
Brief Title: Ginger Capsules for the Chronic Treatment of Obesity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Antonio L Teixeira Jr, MD, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 30409114.8.0000.5149
Record Dates: First submitted 2016-02-05; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
Keywords: ginger obesity; ginger inflammation; treatment of obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Conventional treatment (restrictive diet) plus capsules of 200 mg of cellulose (placebo) to be taken three times a day for six months.
  Interventions: Dietary Supplement: Placebo
- Ginger group (Experimental): Conventional treatment (restrictive diet) plus capsules of 200 mg of dry extract of ginger (5% active ingredient) to be taken three times a day for six months.
  Interventions: Dietary Supplement: Dry extract of ginger

INTERVENTIONS:
Dietary Supplement: Dry extract of ginger — Restrictive diet plus three capsules of 200 mg of dry extract of ginger (5% active ingredient) to be taken three times a day for six months.
  Arms: Ginger group
Dietary Supplement: Placebo — Restrictive diet plus three capsules of 200 mg of cellulose to be taken three times a day for six months.
  Arms: Placebo

SUMMARY:
Regarding its complex pathogenesis and clinic-epidemiological meaning, different strategies are needed for the treatment of obesity. Ginger is the rhizome of a plant with thermogenic and anti-inflammatory effects, and may be a promising alternative as add-on strategy in the treatment for obesity. The primary objective of the current study is to assess whether consumption of ginger as an add-on strategy to restrictive diet is effective to reduce fat body percentage, increase basal metabolic rate and improve loss weight.

The secondary objectives are:

* to assess the effect of nutritional intervention in quality of diet and weight loss.
* to evaluate the effect of ginger on behavioral symptoms and peripheral biomarkers in overweight subjects.

DETAILED DESCRIPTION:
Overweight individuals will be interviewed at baseline and after 30, 60, 90, 120, 150 and 180 days from baseline. The following measures will be assessed: body composition (fat body% and free fat body%), anthropometric measures (height, weight, body mass index, waist circumference and abdominal circumference), blood pressure, basal metabolic rate, behavioral symptoms, binge eating (binge eating scale) and peripheral biomarkers. Behavioral symptoms will be assessed using the following self-reported questionnaires: Beck Depression Inventory (depression symptoms), Beck Anxiety Inventory (anxiety symptoms), Medical Outcomes Study 36 - Item Short - Form Health Survey (quality of life) and Perceived Stress Scale (stress).

Enrolled participants will receive restrictive diet calculated on individual requirements aiming at the loss from two to four kilogram per month in addition to capsules of ginger or placebo, as follows:

* Group 1 will receive vials containing 90 capsules of 200mg of dry extract of ginger (5% active ingredient) to be taken three times a day for six months in addition to restrictive diet.
* Group 2 will receive vials containing 90 capsules of 200mg of placebo (cellulose) to be taken three times a day for six months in addition to restrictive diet.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-60 years old;
* Body mass index 25-35 kg/m².

Exclusion Criteria:

* Pregnant or lactating women;
* Abuse of alcohol or drugs;
* Hypersensitivity to ginger;
* Other endocrine disease;
* Women in use of insulin or anti-inflammatory and antidepressants drugs.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change in basal metabolic rate. | Baseline and 30, 60, 90, 120, 150 and 180 days
  Ginger effect in basal metabolic rate will be measured by calorimetry.
Change in body fat percentage. | Baseline and 30, 60, 90, 120, 150 and 180 days
  Ginger effect in body fat percentage will be measured by bioimpedance.

SECONDARY OUTCOMES:
Changes in serum levels of inflammatory mediators | Baseline and 30, 60, 90, 120, 150 and 180 days
  Nutritional effect in the levels of Interleukin-1, interleukin-6 and interleukin-10, tumor necrosis factor and protein C reactive.
Change in depressive symptoms. | Baseline and 30, 60, 90, 120, 150 and 180 days
  Nutritional effect in depressive symptoms will be measured by the Beck Depression Inventory.
Change in anxiety symptoms. | Baseline and 30, 60, 90, 120, 150 and 180 days
  Nutritional effect in anxiety symptoms will be measured by the Beck Anxiety Inventory.
Change in quality of life. | Baseline and 30, 60, 90, 120, 150 and 180 days
  Nutritional effect in quality of life will be measured by Medical Outcomes Study 36 - Item Short - Form Health Survey.
Change in perceived stress. | Baseline and 30, 60, 90, 120, 150 and 180 days
  Nutritional effect in perceived stress will be measured by the Perceived Stress Scale.
Change in quality of diet. | Baseline and 30, 60, 90, 120, 150 and 180 days
  Nutritional effect in quality of diet will be measured by the Healthy Eating Index-10.
Changes in serum levels of neurotrophic factors | Baseline and 30, 60, 90, 120, 150 and 180 days
  Nutritional effect in the serum levels of Brain-derived neurotrophic factor, glial-derived neurotrophic factor and neurotrophin-3 and neurotrophin 4/5.

CONTACTS AND LOCATIONS:
Overall Officials: Adaliene VM Ferreira, PhD, Study Director — Federal University of Minas Gerais; Nayara M Monteze, Ma, Study Chair — Federal University of Minas Gerais; Antônio L Teixeira, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Hospital das Clínicas, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Reedt Dortland AK, Giltay EJ, van Veen T, Zitman FG, Penninx BW. Longitudinal relationship of depressive and anxiety symptoms with dyslipidemia and abdominal obesity. Psychosom Med. 2013 Jan;75(1):83-9. doi: 10.1097/PSY.0b013e318274d30f. Epub 2012 Nov 28. PMID 23197842
- [Background] Atashak S, Peeri M, Azarbayjani MA, Stannard SR, Haghighi MM. Obesity-related cardiovascular risk factors after long- term resistance training and ginger supplementation. J Sports Sci Med. 2011 Dec 1;10(4):685-91. eCollection 2011. PMID 24149559
- [Background] Chrubasik S, Pittler MH, Roufogalis BD. Zingiberis rhizoma: a comprehensive review on the ginger effect and efficacy profiles. Phytomedicine. 2005 Sep;12(9):684-701. doi: 10.1016/j.phymed.2004.07.009. PMID 16194058
- [Background] Gregersen NT, Belza A, Jensen MG, Ritz C, Bitz C, Hels O, Frandsen E, Mela DJ, Astrup A. Acute effects of mustard, horseradish, black pepper and ginger on energy expenditure, appetite, ad libitum energy intake and energy balance in human subjects. Br J Nutr. 2013 Feb 14;109(3):556-63. doi: 10.1017/S0007114512001201. Epub 2012 Jul 5. PMID 23021155
- [Background] Saravanan G, Ponmurugan P, Deepa MA, Senthilkumar B. Anti-obesity action of gingerol: effect on lipid profile, insulin, leptin, amylase and lipase in male obese rats induced by a high-fat diet. J Sci Food Agric. 2014 Nov;94(14):2972-7. doi: 10.1002/jsfa.6642. Epub 2014 Apr 7. PMID 24615565